CLINICAL TRIAL: NCT02861547
Title: Development and Validation of a Prognostic Score for Early Death in Head Injury Patients in the Traumatic Brain Injury Intensive Care Unit of Dijon CHU
Brief Title: Development and Validation of a Prognostic Score for Early Death in Head Injury Patients.
Acronym: SCORE TC
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Centre Hospitalier Universitaire Dijon (Other)
Responsible Party: Sponsor
Other Study IDs: MIREK 2015
Record Dates: First submitted 2016-08-05; First posted 2016-08-10 (Estimated); Last update posted 2016-08-10 (Estimated); Status verified 2016-07

CONDITIONS: Traumatic Brain Injury
MeSH Terms: conditions — Brain Injuries, Traumatic | interventions — Death Domain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

GROUPS / COHORTS (1):
- Traumatic brain injury
  Interventions: Other: death

INTERVENTIONS:
Other: death

SUMMARY:
Traumatic brain injury (TBI) is a serious condition with high morbidity and mortality. The Glasgow score alone, assessed at the initial phase, is not enough to determine the prognosis.

The aim of this study is to define and to evaluate a prognostic score for early death based on clinical and CT-scan findings in an observational retrospective derivation cohort of patients hospitalized for traumatic brain injury.

This cohort will allow us to carry out a uni- and then multi-variate analysis so as to create a prognostic score for early death.

We will subsequently test this score in a prospective validation cohort.

ELIGIBILITY:
Inclusion Criteria:

Traumatic brain injury (PMSI code (Programme Médicalisation des Systèmes d'Information) S 06.70 and S 06.71) Age>14 years Surviving more than 6h after the trauma Hospitalized in the traumatic brain injury intensive care unit and managed in accordance with international guidelines Who underwent a cerebral CT-scan

Exclusion Criteria:

Ongoing treatment with anticoagulants or antiplatelets Pregnant women Persons without national health insurance cover Children less than 15 years old Under guardianship.

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients hospitalisés pour traumatic brain injury
Sampling Method: Non-Probability Sample
Enrollment: 355 (Estimated)
Dates: Start 2015-05; Primary Completion 2017-05 (Estimated)

PRIMARY OUTCOMES:
Early death | Through the study completion up to 2 years

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Dijon Bourgogne, Dijon, France